CLINICAL TRIAL: NCT00796094
Title: Elasticity Imaging of Soft Tissues
Brief Title: Imaging of Soft Tissues
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yoav Morag, MD, Associate Professor of Radiology, University of Michigan
Other Study IDs: HUM 20943
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Soft Tissue Injury
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Evaluation of tissue elasticity: Evaluate the potential importance of tissue elasticity in the assessment soft tissue structures.
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Sonoelastrography is an ultrasound examination that can determine the elasticity of soft tissue. This examination takes approximately 10 minutes to complete.

SUMMARY:
The purpose of this study is to evaluate the potential importance of tissue elasticity in the assessment of soft tissues including muscles, tendons and ligaments and other soft tissue structures.

The evaluation of tissue elasticity (easily stretched or moveable) may assist in assessment of various soft tissue structures, such as fatty atrophy of muscles, tendon/ligamentous injury and healing and other soft tissue structures.

DETAILED DESCRIPTION:
This is a prospective study that will recruit males and females 18 years of age and older who present to the department for a clinically indicated ultrasound of a superficial soft tissue abnormality with prior or following MRI / CT assessment ordered for clinical purposes.

The elasticity properties of tissues depend on their molecular building blocks and on the organization of these blocks. Injuries, disease etc are known to be associated with changes in tissue elasticity. Little research has been done on the potential of sonoelastographic (elasticity ultrasound imaging) assessment of normal, injured or healing muscles, tendons or ligaments.

Elasticity changes in muscle, ligaments and tendons following injury may have implication on the choice of treatment and help in determine how the length of time needed to heal from an injury.

Stiffness/elasticity of the tissue can be assessed by mechanical excitation with measurement of resultant tissue motion. Reconstruction of the elastic deformability (strain imaging) in real time ultrasound is known as sonoelastography.

Elasticity ultrasound imaging will be performed on the area being evaluated clinically.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who present for a clinically ordered ultrasound for evaluation of a soft tissue abnormality.

Exclusion Criteria:

* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and non pregnant females with soft tissue abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To assess the potential importance of Sonoelastography in evaluating tissue injury or abnormalities of soft tissues. | hours

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Morag, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided